CLINICAL TRIAL: NCT04379674
Title: Effect of Kinesiotaping in Different Directions on Muscle Endurance in Healthy Individuals
Brief Title: Effect of Kinesiotaping in Different Directions on Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Hilal UZUNLAR, Graduate Student at Mugla Sıtkı Koçman University and Research Assistant at Hitit University, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 190079
Record Dates: First submitted 2020-05-06; First posted 2020-05-07 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: KINESIOTAPING
Keywords: KINESIOTAPING; FACILITATION; INHIBITION; ENDURANCE; HEALTHY INDIVIDUAL
MeSH Terms: conditions — Inhibition, Psychological

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Grup 1- Facilitation (Experimental): It consists of cases that start with the taping of the facilitation.
  Interventions: Other: FACILITATION TAPING; Other: INHIBITION TAPING; Other: PLACEBO TAPING
- Grup 2- İnhibition (Experimental): It consists of cases that start with the taping of the inhibition.
  Interventions: Other: FACILITATION TAPING; Other: INHIBITION TAPING; Other: PLACEBO TAPING
- Grup 3- Plasebo (Placebo Comparator): It consists of cases that start with the taping of the placebo.
  Interventions: Other: FACILITATION TAPING; Other: INHIBITION TAPING; Other: PLACEBO TAPING

INTERVENTIONS:
Other: FACILITATION TAPING — The muscle technique, which is a kinesio tape technique, will be used in the biceps brachii muscle. Taping was done with 25% tension with Y tape from the origin to insertion of the muscle.
Other: INHIBITION TAPING — The muscle technique, which is a kinesio tape technique, will be used in the biceps braki muscle. Taping was done with 25% tension with Y tape from the insertio to origo of the muscle.
Other: PLACEBO TAPING — Unlike Kinesio taping muscle technique, it was performed with horizontal taping on the muscle. The ends of the kinesio tapes will be applied tension-free without overlapping with I tape.

SUMMARY:
The study was conducted to investigate the effects of different Kinesio taping directions on dynamic muscle endurance. This randomized, double-blind, crossover study was implemented on 27 healthy male subjects. Before the study, personal and demographic information of the volunteers were recorded and muscle strength was evaluated in the biceps curl position with 1 maximum repetition technique. One week after this first evaluation muscle endurance was evaluated by counting the accurate elbow flexions completed in biceps curl position with 80% weight of 1 maximum repetition recorded in the first evaluation. Following this second evaluation facilitation, inhibition, and placebo tapings were applied to all the 27 subjects who were randomly assigned into 3 groups sequentially with an interval of two days. The sequence of taping technique to be used for the groups were also randomly determined and applied to the M. Biceps Brachii and muscle endurance was evaluated with the same method half-hour after the tape was applied. All the evaluations were performed by the same evaluator who was blind to the taping technique.

DETAILED DESCRIPTION:
Facilitation taping was applied from the origins of the muscle to the insertion. Inhibition taping was applied from the insertio of the muscle to the origin. Facilitation taping and inhibition taping was applied on the target tissue with 25% tension. Y-band was used during facilitation taping and inhibition taping. It was applied to individuals with shoulder mild abduction, external rotation, elbow extension and supination position. Placebo taping was applied while in a resting position. In placebo taping, it was applied using two I bands in horizontal direction. In placebo taping, no tension was applied to the tapes. Evaluations were made while the subjects were standing. The biceps curl exercise position starts with the palms facing the trunk. Elbow flexion is completed by making full range of motion. The cases were randomized into 3 groups: group-1 facilitation taping, group-2 inhibition taping and group-3 placebo taping.The treatment sequence to be applied to the patients was determined by randomization. Facilitation, inhibition and placebo banding were applied to the patients, respectively. Accordingly, inhibition and placebo taping was applied to the cases that started with the facilitation taping. Placebo and facilitation banding were applied to the patients that started with inhibition banding, respectively. Facilitation and inhibition banding was applied to the cases that started with placebo banding, respectively. During the evaluation, banding application was kept by wearing plenty of clothes. Evaluators and subjects participating in the study did not have knowledge and experience about the taping method.

ELIGIBILITY:
Inclusion Criteria:

* Being a male university student over the age of 18
* Volunteering for the study
* Fiiling out the informed consent form not having the knowledge and experience about kinesiotaping before

Exclusion Criteria:

* Anabolic agent users
* Having any neurological disease or systemic disease
* Having undergone spine and upper extremity surgery
* Skin sensitivity to elastic banding
* Open wound, ulser, fungal infection in the area to be taped
* Exposure to upper extremity and/or spinal injury in the past 6 months
* To have used alcohol, caffeine-containing substances and pain medication in the last 24 hours before the evaluation.
* To have been involved in physical activity and / or activities in the last 48 hours prior to the evaluation, other than routine work, that will tire the upper limbs.

Ages: 18 Years to 27 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 27 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2019-05-13 (Actual); Study Completion 2019-07-12 (Actual)

PRIMARY OUTCOMES:
Number of Elbow Flexion | 2 minutes
  Muscle endurance was found by recording the number of elbow flexions performed within 1 minute in the biceps curl exercise position against moderate violence at the rate of 80% of 1 maximum repetition. Facilitation taping, inhibition taping and placebo taping were applied to 27 subjects randomized to 3 groups at two consecutive day intervals. The order of taping was also determined by randomization method and performed on the biceps braki muscle in the dominant limb of the subjects, and muscle endurance was evaluated half an hour after taping.

OTHER OUTCOMES:
Maximum of 1 Repetition (1-MT) | 10 minutes
  Muscle strength was found with a maximum of 1 repetition (1-MT) in the biceps curl exercise position. The subjects were asked to perform the movement against resistance with the greatest weight predicted during this evaluation position. When he was able to repeat the movement a second time or more, we continued by adding 5 kg, 3 kg, 2 kg or 1 kg weights, respectively. 1-MT was found by giving 1 minute rest intervals between repeated trials.

CONTACTS AND LOCATIONS:
Locations (1):
- Mugla Sıtkı Kocman University Health Sciences Faculty, Muğla, Turkey (Türkiye)